CLINICAL TRIAL: NCT00711906
Title: The Role of Daily Co-trimoxazole Prophylaxis For Prevention of Malaria And Its Effects in Pregnancy
Brief Title: Daily Co-trimoxazole Prophylaxis to Prevent Malaria in Pregnancy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Malaria prev. fell in the study area, so we cannot evaluate the primary endpoint
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Tropical Diseases Research Centre, Zambia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ITMP0108
Record Dates: First submitted 2008-07-08; First posted 2008-07-09 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Malaria in Pregnancy
Keywords: Malaria; Pregnancy; HIV; Intermittent Preventive Treatment; Safety; Efficacy
MeSH Terms: conditions — Malaria | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): HIV-negative women taking CTX as chemoprophylaxis
  Interventions: Drug: Cotrimoxazole
- 2 (Active Comparator): HIV-negative women taking SP as IPT
  Interventions: Drug: Sulfadoxine-pyrimethamine
- 3 (Experimental): HIV-positive women (CD4> 200) taking CTX as chemoprophylaxis
  Interventions: Drug: Cotrimoxazole
- 4 (Active Comparator): HIV-positive women (CD4 > 200) taking SP as IPT
  Interventions: Drug: Sulfadoxine-pyrimethamine

INTERVENTIONS:
Drug: Cotrimoxazole — Cotrimoxazole
  Other Names: CTX; Bactrim
  Arms: 1; 3
Drug: Sulfadoxine-pyrimethamine — Sulfadoxine-pyrimethamine
  Other Names: SP; Fansidar
  Arms: 2; 4

SUMMARY:
Malaria is a major contributor of disease burden in Sub-Saharan Africa, and pregnant women and children are the most vulnerable population. Malaria in pregnancy increases the risks of abortion, prematurity, maternal anaemia, low birth weight (LBW), perinatal, neonatal and infant mortality. For prevention and control of malaria in pregnancy, Intermittent Preventive Treatment (IPT), insecticide treated nets (ITNs) and case management for malaria and anemia are recommended.

HIV infection in pregnancy increases the risk of malaria, LBW, post-natal mortality and also of anaemia. In pregnant women, HIV infection decreases the efficacy of IPT with the medicine sulfadoxine-pyrimethamine (SP), which is the only treatment with proven efficacy and safety in IPT and is recommended by the World Health Organization (WHO). Unfortunately, there is a documented increase of resistance to SP, so cotrimoxazole (CTX) could be an alternative: many studies in Zambia and Uganda demonstrated that it reduces mortality and morbidity in HIV infected persons, and CTX prophylaxis significantly improves birth outcomes in immuno-suppressed HIV women. Unfortunately, there is not yet information on its effectiveness for preventing placental malaria infection, maternal anaemia and LBW. Thus in this study, we aim to establish the safety and efficacy of daily CTX in preventing malaria infection during pregnancy and its consequences, both in HIV infected and non-infected pregnant women. This information is urgently needed to assist to issue guidelines on IPT in pregnancy.

DETAILED DESCRIPTION:
Malaria is a major contributor of disease burden in Sub-Saharan Africa, with pregnant women and children being the most vulnerable population. P. falciparum infection in pregnancy leads to parasite sequestration in placental vascular space, with increased risks of abortion, stillbirth, prematurity, intrauterine growth retardation, maternal anaemia, low birth weight (LBW), perinatal, neonatal and infant mortality. In low transmission areas, malaria can evolve towards severe disease with high risk of mortality. In endemic areas, it is still associated with maternal anaemia, LBW and stillbirth. For prevention and control of malaria in pregnancy, WHO recommends Intermittent Preventive Treatment (IPT), insecticide treated nets (ITNs) and case management for malaria and anemia.

HIV in pregnancy increases the risk of malaria, LBW, post-natal mortality and also anaemia, suggesting a synergistic interaction between HIV and malaria.

In pregnant women, HIV-1 infection decreases the efficacy of sulfadoxine-pyrimethamine(SP)IPT, although 2 or more doses in 2nd and 3rd trimesters still reduce peripheral parasitaemia, placental infections and maternal anaemia.

To date, SP is the only treatment with data on efficacy and safety in IPT: WHO recommends at least 2 doses after the first trimester. But there is a documented increase in SP resistance, so cotrimoxazole (CTX) could be an alternative: many studies in Zambia and Uganda demonstrated that it reduces mortality and morbidity in HIV infected individuals, and CTX prophylaxis significantly improves birth outcomes in women with CD4 count <200. Concurrent administration of SP and CTX has been associated with increased incidence of severe adverse reactions in HIV-infected patient.

WHO has promoted CTX as alternative to SP for IPT in immuno-compromised HIV-infected pregnant women. Unfortunately, there is no information on effectiveness of daily CTX for preventing placental malaria infection, maternal anaemia and LBW. In the past, CTX has been used to treat malaria in children and daily use of CTX by non-pregnant HIV-infected adults has been associated with a 70% reductions of the incidence of clinical malaria.

In this study, we will target both HIV infected and non-infected pregnant women with CD4≥ 200/µL, with the aim to establish the safety and efficacy of daily CTX in preventing malaria infection during pregnancy and its consequences, by assuming that CTX is not inferior to SP in reducing placental parasitaemia: such information is urgently needed to assist to issue guidelines on IPT in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pregnancy (through palpable fundus and/ or positive pregnancy test)
* Gestational age between 16 and 28 weeks.
* Informed consent by patient (or parent/ guardian if patient is less than 18 years of age)
* No symptoms consistent with malaria
* Willingness to deliver at the health facility
* Willingness to adhere to all requirements of the study (including HIV-1 testing)

Exclusion Criteria:

* History of allergy to study drugs, or previous history of allergy to sulpha drugs
* History or presence of major illnesses likely to influence pregnancy outcome including diabetes mellitus, severe renal or heart disease, or active tuberculosis, prior to randomization;
* Any significant illness that requires hospitalization;
* Intent to move out of the study catchment's area before delivery or deliver at relative's home out of the catchment's area;
* Prior enrolment in the study or concurrent enrolment in another study
* Severe anaemia (Hb<7 g/dl)
* Previous history of unfavourable pregnancy outcome: pre-eclampsia, caesarean section, stillbirth.
* Being HIV infected and already receiving CTX prophylaxis or ARV treatment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To test the hypothesis that co-trimoxazole prophylaxis is not inferior to SP intermittent preventive treatment in preventing placental malaria. | Pregnancy

SECONDARY OUTCOMES:
To evaluate efficacy of CTX prophylaxis in preventing malaria peripheral parasitaemia. | Pregnancy
To evaluate efficacy of CTX prophylaxis in preventing perinatal mortality and in improving birth weight | At birth
To establish the safety of CTX prophylaxis on the offspring by measuring the gestational age at delivery and birth weight. | At birth
To compare the efficacy profile of CTX prophylaxis to that of SP intermittent preventive treatment. | Pregnancy
To compare the safety profile of CTX prophylaxis to that of SP intermittent preventive treatment. | Pregnancy
Spontaneous abortion | </=28 weeks gestation
Pre-term delivery | <37 completed weeks
Neonatal mortality | Within 28 days after birth
Maternal mortality | Up to 6 weeks following delivery
Major and minor birth defects | At birth and up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christine Manyando, MD, Principal Investigator — Tropical Diseases Research Centre; Jean-Pierre Van geertruyden, MD PhD, Study Director — Institute of Tropical Medicine
Locations (2):
- Zambia (2):
  - Choma hospital, Choma
  - Shampande Clinic, Shampande

REFERENCES:
- [Derived] Pons-Duran C, Wassenaar MJ, Yovo KE, Marin-Carballo C, Briand V, Gonzalez R. Intermittent preventive treatment regimens for malaria in HIV-positive pregnant women. Cochrane Database Syst Rev. 2024 Sep 26;9(9):CD006689. doi: 10.1002/14651858.CD006689.pub3. PMID 39324693
- [Derived] Manyando C, Njunju EM, Mwakazanga D, Chongwe G, Mkandawire R, Champo D, Mulenga M, De Crop M, Claeys Y, Ravinetto RM, van Overmeir C, Alessandro UD, Van Geertruyden JP. Safety of daily co-trimoxazole in pregnancy in an area of changing malaria epidemiology: a phase 3b randomized controlled clinical trial. PLoS One. 2014 May 15;9(5):e96017. doi: 10.1371/journal.pone.0096017. eCollection 2014. PMID 24830749
- See also: study results — http://www.plosone.org/article/info%3Adoi%2F10.1371%2Fjournal.pone.0096017;jsessionid=5BFAF926D82FA94E2B41060D2FFBE596